CLINICAL TRIAL: NCT00357253
Title: A Phase I Trial of Capecitabine Rapidly Disintegrating Tablets and Concomitant Radiation Therapy in Children With Newly Diagnosed Brainstem Gliomas and High Grade Gliomas
Brief Title: Capecitabine and Radiation Therapy in Treating Young Patients With Newly Diagnosed, Nonmetastatic Brain Stem Glioma or High-Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000484429; U01CA081457 (NIH); PBTC-021
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma; childhood high-grade cerebral astrocytoma; untreated childhood cerebellar astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine — This is a dose escalation study. 375, 500, 650, or 850 mg/m2 capecitabine RDT is given orally daily in two divided doses approximately 12 hours apart beginning at the start of radiation therapy and continuing for 9 weeks. After a two week break, patients receive twice daily oral capecitabine, either 900 mg/m2 or 1250 mg/m2, approximately 12 hours apart for 14 days followed by a 7-day rest period for a total of 3 courses.
  Other Names: Xeloda
Radiation: radiation therapy — Participants receive local radiation once daily, 5 days/week for 9 weeks for a total dose of 5580 cGy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Capecitabine may make tumor cells more sensitive to radiation therapy. Giving capecitabine together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of capecitabine when given together with radiation therapy in treating young patients with newly diagnosed, nonmetastatic brain stem glioma or high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the maximum tolerated dose of capecitabine rapidly disintegrating tablets (RDT) administered concurrently with radiotherapy in young patients with newly diagnosed, nondisseminated intrinsic brain stem glioma or high-grade glioma.
* Describe the dose-limiting toxicity in patients treated with this regimen.

Secondary

* Describe the safety profile of this regimen.
* Characterize the pharmacokinetics of capecitabine RDT in these patients.
* Explore the exposure-response relationship for measures of safety and effectiveness using pharmacokinetic and pharmacodynamic models.
* Describe the antitumor activity of this regimen observed in these patients.
* Estimate distributions of progression-free survival and survival in patients treated with this regimen.
* Characterize radiographic changes in tumor, using MRI, perfusion and diffusion MRI, and positron emission tomography (PET) scans, in patients treated with this regimen.

OUTLINE: This a multicenter, dose-escalation study of capecitabine rapidly disintegrating tablets (RDT).

Patients undergo radiotherapy once daily, 5 days a week, for approximately 6 weeks. Beginning within 24 hours of starting radiotherapy, patients also receive oral capecitabine RDT twice daily on days 1-21. Treatment with capecitabine RDT repeats every 21 days for 3 courses.

Cohorts of 3-6 patients receive escalating doses of capecitabine RDT until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Beginning in week 12, patients receive capecitabine RDT at a fixed dose twice daily on days 1-14. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during course 1 for pharmacokinetic correlative studies. Patients also undergo MRI, and rapid perfusion/diffusion MRI at baseline and periodically during study for radiographic correlative studies.

After completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following newly diagnosed, nondisseminated brain tumors:

  * Intrinsic infiltrating brain stem glioma

    * Histopathologic diagnosis not required
  * Histopathologically confirmed high-grade glioma, meeting all of the following criteria:

    * Underwent prior definitive surgery ≤ 28 days ago with incompletely resected disease
    * Any of the following subtypes allowed:

      * Anaplastic astrocytoma
      * Glioblastoma multiforme
      * Other high-grade glioma
* No anaplastic oligodendroglioma

PATIENT CHARACTERISTICS:

* Karnofsky performance scale (PS) 50-100% (if > 16 years of age) or Lansky PS 50-100% (if ≤ 16 years of age)
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 8 g/dL (transfusion independent)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR creatinine based on age as follows:

  * No more than 0.8 mg/dL (for patients 5 years of age and under)
  * No more than 1 mg/dL (for patients 6-10 years of age)
  * No more than 1.2 mg/dL (for patients 11-15 years of age)
  * No more than 1.5 mg/dL (for patients over 15 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No significant cardiac, hepatic, gastrointestinal, renal, pulmonary, or other systemic disease
* No known hypersensitivity to capecitabine or any of its components
* No known dihydropyrimidine dehydrogenase (DPD) deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior dexamethasone and/or surgery allowed
* No prior chemotherapy, radiotherapy, immunotherapy, or bone marrow transplantation
* No other concurrent anticancer or experimental drug therapies or agents
* No concurrent warfarin or sorivudine or its chemically related analogues (e.g., brivudine)

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of capecitabine rapidly disintegrating tablets (RDT) in combination with radiotherapy | First 11 weeks of therapy
Dose-limiting toxicity | First 11 weeks of therapy

SECONDARY OUTCOMES:
Pharmacokinetics of capecitabine RDT measured periodically during course 1 | Day 1 and Day 14 of therapy
Tumor response | From day 1 of treatment until off study
  Brain imaging to assess tumor response to the treatment is performed at baseline, week 11, end of course 6, and then every 3 months for two years.
Survival | From initiation of treatment until death or off study
Radiographic changes in gliomas as measured by MRI, magnetic resonance spectroscopy (MRS), perfusion and diffusion MRI | Baseline, week 11, then every 3 months for 2 years or until off study

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Blaney, MD, Study Chair — Texas Children's Cancer Center
Locations (12):
- United States (12):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington